CLINICAL TRIAL: NCT01092910
Title: Esteem Totally Implantable Hearing System Clinical Trial U.S. Pivotal Trial
Brief Title: Esteem Totally Implantable Hearing System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Envoy Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0204
Record Dates: First submitted 2010-03-19; First posted 2010-03-25 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2016-01

CONDITIONS: Mild to Severe Sensorineural Hearing Loss
Keywords: Sensorineural; Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Esteem Implant (Experimental): Subjects are implanted with the Esteem Totally Implantable Hearing System
  Interventions: Device: Esteem Totally Implantable Hearing System

INTERVENTIONS:
Device: Esteem Totally Implantable Hearing System — The Esteem System is a totally implantable hearing system designed to improve hearing in adult subjects suffering from mild to severe hearing loss that is sensorineural in origin.

SUMMARY:
To evaluate the safety and efficacy of the Esteem Totally Implantable Hearing System in subjects suffering from mild to severe hearing loss.

DETAILED DESCRIPTION:
Title: Esteem® Totally Implantable Hearing System Clinical Trial

Purpose: To evaluate the safety and efficacy of the Esteem® Totally Implantable Hearing System (hereafter called the Esteem® System) in subjects suffering from mild to severe hearing loss.

Trial Design: This pivotal trial is designed as a prospective, multi-center, non-randomized, clinical trial to evaluate the safety and efficacy of the Esteem® System. For this trial the subject will act as his or her own control.

This trial has been designed to meet the United States' regulatory requirements.

Enrollment Size: It is currently estimated that 50-60 subjects will be enrolled in this trial.

Subject Population: Adult subjects who have mild to severe sensorineural hearing loss, have a healthy middle ear, have a speech discrimination score of equal to or better than 40%, and have previously worn a hearing aid for a minimum of 3 months with an average daily use rate of at least 4 hours are eligible for inclusion in the trial. See detailed inclusion/exclusion criteria for specifics.

Primary Objectives:

1. To demonstrate that the Esteem® System improves the speech threshold of sensitivity for hearing and identifying speech signals as well as or better than the pre-implant hearing aid (aided condition).

   Endpoint: Comparison of the speech reception threshold (SRT) using the Esteem® System (4 months post activation) as compared to the pre-implant aided condition.
2. To demonstrate that the Esteem® System at the 4 months post- activation visit is as effective as or better than the hearing aid for improving speech discrimination (intelligibility) as shown by the word recognition score at 50 dB.

   Endpoint: Comparison of the word recognition score using the Esteem® at 4 months post-activation compared to the pre-implant aided condition.
3. To determine the incidence of Serious Adverse Device Effects (SADE) and the incidence rate of device failures and replacements.

   Endpoint: The analysis of the incidence of SADEs and device failures and replacements at each follow-up.
4. To demonstrate that the subjects' cochlear function remains unchanged with the Esteem® System as shown by comparison of the subjects' pre-implant baseline bone conduction threshold versus the subjects' 4 month post-activation visit bone conduction threshold.

Endpoint: Comparison of bone conduction threshold (BC) using forehead placement at 4 months post activation compared to the pre-implant BC threshold.

Secondary Objectives:

1. To demonstrate that the Esteem® System at the 4 months post activation visit improves the 3-frequency (500, 1000, and 2000 Hz) pure tone average (PTA) when compared to the baseline unaided condition.
2. To demonstrate that the Esteem® System at the 4 months post-activation visit is as effective as or better than the hearing aid for improving speech discrimination (intelligibility) as shown by the QuickSIN (speech in noise) test results.
3. To show that the Esteem® System improves Quality-of-Life when compared to the baseline aided condition as shown by APHAB results.
4. To gather subject feedback and comments on the use of the Esteem® System relative to the pre-implant hearing aid (aided condition) as shown by the Esteem® Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years old
* Subject understands the nature of the procedure and has signed the Subject Informed Consent Form prior to the procedure
* Subject is willing and able to comply with specified follow-up evaluations and understands the audiological test procedures and use of the Esteem System.
* Subject has mild to severe sensorineural hearing loss between 500 and 4000 Hz in the ear to be implanted with pure tone air-conduction threshold levels within the limits of a Hearing Aid (HA) as follow:

Freq (Hz) 500 1000 2000 3000 4000 LL* (dB HL) 30 35 35 35 35 UL* (dB HL) 100 100 100 100 100

*LL = Lower Level; UL = Upper Level

* Subject's air-bone gap is no greater than 10 dB at 4 of the 5 following frequencies: 500, 1000, 2000, 3000 and 4000 Hz.
* Subject has an unaided maximum word recognition score of greater than or equal to 60% with recorded delivery using a phonetically balanced word list at SRT + 40 dB or at maximum tolerable presentation level.
* Subject is a current user of a properly functioning and appropriately fit hearing aid. This is defined as the subject has used this aid for at least four (4) hours (average) per day (in the ear to be implanted) for at least three (3) months for a new aid or one (1) month for an adjusted aid.
* Subject's hearing aid, in the ear to be implanted, shall appropriately fit optimally.
* Subject has normally functioning eustachian tube
* Subject has normal tympanic membrane
* Subject has a normal middle ear anatomy
* Subject has adequate space for Esteem System implant determined via fine cut temporal bone CT scan
* Subject is a native speaker of the English language.
* Subject is a hearing aid user in the ear to be implanted.

Exclusion Criteria:

* Subject has a history of post-adolescent chronic middle ear infections, inner ear disorders or recurring vertigo requiring treatment, disorders such as mastoiditis, Hydrops or Meniere's syndrome or disease
* Subject has a history of otitis externa or eczema for the outer ear canal and the investigator believes this will affect the Esteem System implantation
* Subject has cholesteatoma or destructive middle ear disease
* Subject has life expectancy of two (2) years due to other medical conditions
* Subject has retrocochlear or central auditory disorders
* Subject is known to be suffering from any psychological, developmental, physical, or emotional disorder that the investigator feels would interfere with the surgery or follow-up testing
* Subject has a known history of fluctuating air conduction and/or bone conduction hearing loss over a one-year period of 15 dB in either direction at 2 or more frequencies (from 500 - 4000 Hz)
* Subject has sudden hearing loss due to unknown cause
* Subject has a history of disabling tinnitus, defined as tinnitus which required treatment.
* Subject is unable to adequately perform audiological testing
* Subject has a medical condition or undergoing a treatment that may affect healing and the investigator does not believe the subject is a good candidate for the trial.
* Subject has diabetes that is not well controlled with medication or diet and the investigator does not believe in his best medical judgment that the subject would be a good candidate for the trial
* Subject is pregnant at the time of device implant
* Subject has a history of keloid formation
* Subject has known hypersensitivity to silicone rubber, polyurethane, stainless steel, titanium and/or gold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A. Shohet, M.D., Principal Investigator; Eric M. Kraus, M.D., M.S., Principal Investigator — F.A.C.S.; Peter J. Catalano, M.D., Principal Investigator — F.A.C.S.
Locations (5):
- United States (5):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Shohet Ear Associates, Newport Beach, California
  - Lahey Clinic, Inc., Burlington, Massachusetts
  - Surgical Care Affiliates, Greensboro, North Carolina
  - The Ear Center of Greensboro, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Envoy Medical Corporation Official Web Site — http://www.envoymedical.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at three different sites:
  The Ear Center of Greensboro Greensboro, NC 27401
  Shohet Ear Associates Medical Group, Inc. Newport Beach, CA 92663
  Lahey Clinic Burlington, MA 01805
Period: Overall Study
Arm/Group | Esteem Implant
Started | 57
4 Month Follow-up | 54
10 Month Follow-up | 52
Completed | 52
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Esteem Implant: Subjects implanted with the Esteem Totally Implantable Hearing System
Arm/Group | Esteem Implant
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 56
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: SRT Change
Description: Comparison of the speech reception threshold (SRT) using the Esteem System as compared to the pre-implant aided condition
Time Frame: 4 Months Post Activation
Measure: Mean (Standard Error); unit: dB
Groups:
- Esteem Implant: Subjects implanted with the Esteem Totally Implantable Hearing System
  The Esteem System is a totally implantable hearing system designed to improve hearing in adult subjects suffering from mild to severe hearing loss that is sensorineural in origin.
Arm/Group | Esteem Implant
Number analyzed (Participants) | 54
dB | 10.6 (1.6)

2. Primary Outcome: SRT Change
Description: as for outcome 1
Time Frame: 10 Months Post-Activation
Measure: Mean (Standard Error); unit: dB
Arm/Group | Esteem Implant
Number analyzed (Participants) | 54
dB | 11.4 (1.8)

3. Primary Outcome: Word Recognition Score Change
Description: Comparison of the word recognition score using the Esteem compared to the pre-implant aided condition
Time Frame: 4 Months Post Activation
Measure: Mean (Standard Error); unit: change in % correct
Arm/Group | Esteem Implant
Number analyzed (Participants) | 52
change in % correct | 21.7 (4.2)

4. Primary Outcome: Word Recognition Score Change
Description: Comparison of the word recognition score using the Esteem compared to the pre-implant aided condition
Time Frame: 10 Months Post Activation
Measure: Mean (Standard Error); unit: change in % correct
Arm/Group | Esteem Implant
Number analyzed (Participants) | 52
change in % correct | 19.8 (4.3)

5. Primary Outcome: SADEs
Description: The incidence of Serious Adverse Device Effects (SADE) and the incidence rate of device failures and replacements
Time Frame: 10 Months Post-Activation
Population: Includes all events, cumulatively, from enrollment through 10-month followup
Measure: Number; unit: events
Arm/Group | Esteem Implant
Number analyzed (Participants) | 57
events | 6

6. Primary Outcome: Assessment of Cochlear Function at 4-months and 10-months Post-activation, as Evidenced by Bone-conduction (BC) Thresholds.
Description: Comparison of bone conduction thresholds at the 4-month and 10-month post-activation follow-up, relative to the pre-implant baseline bone conduction thresholds. Lower thresholds represent better (more sensitive) outcomes.
Time Frame: Baseline, 4-, and 10-Months Post-Activation
Population: 4-month and 10-month BC PTA (average 500, 1kHz, 2kHz) compared to baseline BC PTA
Measure: Mean (Standard Error); unit: dB HL
Arm/Group | Esteem Implant
Number analyzed (Participants) | 52
dB HL
  Baseline bone conduction PTA | 55.6 (1.3)
  4 mo. bone conduction PTA | 55.6 (1.2)
  10 mo. bone conduction PTA | 55.3 (1.4)

7. Secondary Outcome: Comparisons of Change in Global Score on Abbreviated Profile of Hearing Aid Benefit (APHAB) at 4 Months and at 10 Months Post-activation, Relative to Pre-implant Baseline Score
Description: To assess whether the Esteem System improves Quality-of-Life, when compared to the baseline aided condition (pre-implant) as shown by the global Abbreviated Profile of Hearing Aid Benefit (APHAB) score. The APHAB is a 24-item self-assessment inventory in which patients report the amount of trouble they are having with communication in various everyday situations using a scale ranging from 0 to 100, with higher scores indicating less difficulty (or increased benefit). The Global Score is the average of 3 subscales.
  Scores reported here are calculated by comparing the patient's reported difficulty in the baseline "unaided" condition with their amount of difficulty when using amplification (hearing aids or implant) -- i.e. Global Scores at pre-implant baseline subtracted from scores at aided baseline and at 4 and 10 months post-implant. Positive numbers denote increased benefit relative to unaided baseline, and the higher the number, the greater the benefit.
Time Frame: 4 and 10 Months Post-Activation
Population: Data from entire subject cohort not available.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Esteem Implant
Number analyzed (Participants) | 46
score on a scale
  Baseline Aided Global Score | 35.0 (2.2)
  4 mo.Global Score with Esteem: number analyzed (Participants) | 43
  4 mo.Global Score with Esteem | 47.9 (3.1)
  10 mo. Global Score with Esteem | 46.6 (3.0)

8. Secondary Outcome: Scores on Esteem Questionnaire
Description: To gain subject feedback on the use of the Esteem System relative to their pre-implant hearing aid (aided condition) as shown by the (unvalidated) Esteem Questionnaire. Subjects completed a 7-item questionnaire rating various subjective attributes concerning their experience with Esteem as compared to their previous hearing aid. Ratings were on a scale of 1 to 5, where 1 is "much worse," 3 is the same and 5 is "much better." Reported here are proportions of participants responding to each score (1 to 5) on the scale, for average scores across all 7 items for each subject.
Time Frame: 4 and 10 Months Post Activation
Measure: Count of Participants; unit: Participants
Arm/Group | Esteem Implant
Number analyzed (Participants) | 49
Participants
  Response "1" - 4 mo average across items | 2
  Response "2" - 4 mo | 5
  Response "3" - 4 mo | 4
  Response "4" - 4 mo | 15
  Response "5" - 4 mo | 23
  Response "1" - 10 mo ave across items | 2
  Response "2" - 10 mo | 3
  Response "3" - 10 mo | 5
  Response "4" - 10 mo | 12
  Response "5" - 10 mo | 24
  Response Missing - 10 mo | 3

9. Secondary Outcome: Change in Pure Tone Average (PTA) at 4 Months, Relative to Baseline Pre-implant
Description: For each subject, the 4-month post-activation Air Conduction PTA (average of thresholds at three frequencies: 500, 1000, and 2000 Hz) was compared to the baseline unaided PTA. A negative mean difference (in dB) from baseline indicates improved hearing sensitivity with the Esteem, relative to baseline.
Time Frame: 4 Months Post Activation
Measure: Mean (Standard Error); unit: dB
Arm/Group | Esteem Implant
Number analyzed (Participants) | 53
dB | -27 (1)

10. Secondary Outcome: Difference in QuickSIN (Quick Speech-In-Noise Test) Score at 4 Months Relative to Baseline Aided Condition
Description: The Quick-SIN is a test of sentence recognition in varying levels of background noise. The score achieved is termed "SNR loss," and a higher score indicates poorer performance on the test. "SNR Loss" is defined as the dB increase in signal-to-noise ratio required by a hearing-impaired person to understand speech in noise, compared to someone with normal hearing. (The range of possible scores is -4.5 to 25.5, with lower scores indicating better performance.) For this study, baseline scores for each subject are subtracted from 4 month scores, providing a difference score. The mean difference across subjects is reported here, with 0 meaning no change and a negative difference indicating better performance with Esteem, compared to the pre-implant aided condition.
Time Frame: 4 Months Post Activation
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Esteem Implant
Number analyzed (Participants) | 53
score on a scale | -1 (1)

ADVERSE EVENTS:
Time Frame: Cumulative through 10 Month Post-Activation
Arm/Group | Esteem Implant
Serious Adverse Events (participants affected / at risk) | 6/57
Other Adverse Events (participants affected / at risk) | 43/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esteem Implant (N=57)
Limited benefit (Ear and labyrinth disorders) | 3 (3)
Incision Breakdown (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain and Facial Weakness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esteem Implant (N=57)
Chorda Tympani/Taste Disturbance (Nervous system disorders) | 23 (24)
Ear effusion/fluid (Ear and labyrinth disorders) | 17 (17)
Tinnitus (Ear and labyrinth disorders) | 8 (9)
Dizziness/vertigo (Ear and labyrinth disorders) | 7 (7)
Incision discomfort/breakdown (Skin and subcutaneous tissue disorders) | 6 (6)
Ear pain (Ear and labyrinth disorders) | 4 (4)
Facial weakness/paralysis (Nervous system disorders) | 4 (4)
Headache/Pain (post-op) (General disorders) | 4 (4)
Ear cracking/roaring (Ear and labyrinth disorders) | 3 (3)
Otitis externa/TM (Ear and labyrinth disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No